CLINICAL TRIAL: NCT01646060
Title: Clinical Evaluation of the Zynex Blood Volume Monitor (CM-1500) in Healthy Male Adult Subjects During a Blood Draw
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZM-11-01
Record Dates: First submitted 2011-11-28; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Blood Loss; Healthy
Keywords: blood; loss; healthy; volume; To evaluate the ability of the Zynex BVM to non-invasively detect blood loss in healthy subjects during a blood draw.
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Draw (Experimental)
  Interventions: Device: CM-1500

INTERVENTIONS:
Device: CM-1500 — Blood Volume Monitor

SUMMARY:
Zynex's blood volume monitor (BVM) is a non-invasive monitoring device to monitor blood volume and blood loss of a patient during surgery, post operatively and/or in recovery. This monitoring device will identify baseline blood volume and relative changes in blood volume using a specific algorithm to compare and review data already monitored during surgery, displaying blood volume and blood loss in real-time.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male, 18-65 years of age
* Subject is suitable for a blood draw of a pint of blood
* Weighs at least 110 pounds

Exclusion Criteria:

* Subject has a heart condition that may interfere with the Zynex CM-1500
* Subject has unstable or untreated heart disease
* Subject has been diagnosed with chronic fatigue syndrome
* Subject is taking coumadin (warfarin), heparin, or other prescription blood thinners for at least 7 days prior to blood draw
* Subject donated blood within 8 weeks prior to blood draw
* Subject has high or low blood pressure on the day of blood draw
* Subject hemoglobin < 12.5 g/dL

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Detect change in blood volume during blood draw | 15-30 minutes

SECONDARY OUTCOMES:
Detect insidious bleeding | 15-30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Moore, MD, Principal Investigator — Rocky Mountain Urgent Care
Locations (1):
- Rocky Mountain Urgent Care, Aurora, Colorado, United States